CLINICAL TRIAL: NCT01683851
Title: Isolite and Dental Treatment Under Conscious Sedation: a Pilot Study to Assess the Upper Airway in a Pediatric Population
Brief Title: Isolite and Dental Treatment Under Conscious Sedation
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Claudia Isabel Contreras, Professor, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC200120233H
Record Dates: First submitted 2012-09-07; First posted 2012-09-12 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Dental Caries
Keywords: pediatric; conscious sedation; mouthpiece; airway; isolite system
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Isolite System — A type of isolation system used in dentistry. It protects soft tissues, and also has a mouth prop, which helps keep mouth open.
  Other Names: Isolite

SUMMARY:
Hypothesis

The use of Isolite® system does not produce upper airway obstruction in the pediatric population during dental treatment with conscious sedation.

Purpose:

Report the changes in airway patency and pediatric patient's behavior when Isolite® system is used for dental treatment with conscious sedation.

Objectives:

1. Determine changes in pulse rate
2. Determine changes in SpO2
3. Recognize breath sound's changes possibly associated with airway blockage
4. Evaluate if the isolite® system is well tolerate by the pediatric population for dental treatment under conscious sedation
5. Relate the use of Isolite® with the frequency of head reposition to open the airway.

DETAILED DESCRIPTION:
Report the changes in airway patency and pediatric patient's behavior when Isolite® system is used for dental treatment with conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I (no systemic disease), ASA II (mid systemic disease-well controlled)
* 4-7 years of age
* Patients English and Spanish speaking

Exclusion Criteria:

* Upper airway infection
* Craniofacial anomalies

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients in need of a sedation dental appointment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Isolite and Dental Treatment Under Conscious Sedation | 120 minutes (sedation appointment time)
  In this study all patients were Mallampati 1 and Brodsky 2. The device comes in 4 sizes: pedo, small, medium and large. The most commonly used was pedo 65% (13) and small 35% (7). Eighty percent (16) of sedations had a satisfactory experience with Isolite ®, Twenty percent (4) had unsatisfactory outcome due to disruptive behavior. Of these 4 cases 2 patients were medicated with meperidine + hydroxyzine and the other 2 with midazolam.
  Fifty percent (8) of the patients successfully treated with Isolite ® experienced snoring and head reposition was performed to open airway. The level of sedation according to the AAPD guidelines was moderate in these events in which snoring occurred. The concentration of nitrous oxide-oxygen was adjusted so that more oxygen was given and the patient would be more alert. No significant changes in SpO2 (mean 99.8) or pulse were observed (mean 90.6).

SECONDARY OUTCOMES:
Isolite and Dental Treatment Under Conscious Sedation | 120 minutes (sedation appointment)
  Finally, it is important to recognize that this is a pilot study with limitations, including:
  1. A small number of participants
  2. No group control
  Therefore, this study's findings need to be tempered by implications contained within these limitations and further research seems indicated.
  Conclusions:
  The results of this pilot study suggest the following conclusions:
  1. Isolite ® may be safely used during pediatric dental treatment under conscious sedation.
  2. The successful use of Isolite ® is related to the patient's behavior. The weakness aspect of Isolite ® is the soft bite block that allows the youngest patients to chew on it.
  Therefore, this study's findings need to be tempered by implications contained within these limitations and further research seems indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia I Contreras, DDS, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - University of Texas Health Science Center-Dental School, San Antonio, Texas
  - University of Texas Health Science Center-Ricardo Salinas Dental Clinic, San Antonio, Texas

REFERENCES:
- [Background] Kameyama A, Asami M, Noro A, Abo H, Hirai Y, Tsunoda M. The effects of three dry-field techniques on intraoral temperature and relative humidity. J Am Dent Assoc. 2011 Mar;142(3):274-80. doi: 10.14219/jada.archive.2011.0166. PMID 21357861
- [Background] Pena BM, Krauss B. Adverse events of procedural sedation and analgesia in a pediatric emergency department. Ann Emerg Med. 1999 Oct;34(4 Pt 1):483-91. doi: 10.1016/s0196-0644(99)80050-x. PMID 10499949
- [Background] Cote CJ, Karl HW, Notterman DA, Weinberg JA, McCloskey C. Adverse sedation events in pediatrics: analysis of medications used for sedation. Pediatrics. 2000 Oct;106(4):633-44. doi: 10.1542/peds.106.4.633. PMID 11015502
- [Background] Cote CJ, Notterman DA, Karl HW, Weinberg JA, McCloskey C. Adverse sedation events in pediatrics: a critical incident analysis of contributing factors. Pediatrics. 2000 Apr;105(4 Pt 1):805-14. doi: 10.1542/peds.105.4.805. PMID 10742324
- [Background] Noro A, Kameyama A, Asami M, Sugiyama T, Morinaga K, Kondou Y, Tsunoda M. Clinical usefulness of "Isolite Plus" for oral environment of Japanese people. Bull Tokyo Dent Coll. 2009 Aug;50(3):149-55. doi: 10.2209/tdcpublication.50.149. PMID 19887758
- [Background] Collette J, Wilson S, Sullivan D. A study of the Isolite system during sealant placement: efficacy and patient acceptance. Pediatr Dent. 2010 Mar-Apr;32(2):146-50. PMID 20483019
- [Background] American Academy on Pediatrics; American Academy on Pediatric Dentistry. Guideline for monitoring and management of pediatric patients during and after sedation for diagnostic and therapeutic procedures. Pediatr Dent. 2008-2009;30(7 Suppl):143-59. PMID 19216414
- [Background] Leelataweedwud P, Vann WF Jr. Adverse events and outcomes of conscious sedation for pediatric patients: study of an oral sedation regimen. J Am Dent Assoc. 2001 Nov;132(11):1531-9; quiz 1596. doi: 10.14219/jada.archive.2001.0086. PMID 11811136
- [Background] Meurice JC, Marc I, Carrier G, Series F. Effects of mouth opening on upper airway collapsibility in normal sleeping subjects. Am J Respir Crit Care Med. 1996 Jan;153(1):255-9. doi: 10.1164/ajrccm.153.1.8542125.
- [Background] MORIKAWA S, SAFAR P, DECARLO J. Influence of the headjaw position upon upper airway patency. Anesthesiology. 1961 Mar-Apr;22:265-70. doi: 10.1097/00000542-196103000-00016. No abstract available. PMID 13772661
- [Background] Verin E, Series F, Locher C, Straus C, Zelter M, Derenne JP, Similowski T. Effects of neck flexion and mouth opening on inspiratory flow dynamics in awake humans. J Appl Physiol (1985). 2002 Jan;92(1):84-92. doi: 10.1152/jappl.2002.92.1.84. PMID 11744646
- [Background] Dickison AE. The normal and abnormal pediatric upper airway. Recognition and management of obstruction. Clin Chest Med. 1987 Dec;8(4):583-96. PMID 3322644
- [Background] Iwatani K, Matsuo K, Kawase S, Wakimoto N, Taguchi A, Ogasawara T. Effects of open mouth and rubber dam on upper airway patency and breathing. Clin Oral Investig. 2013 Jun;17(5):1295-9. doi: 10.1007/s00784-012-0810-5. Epub 2012 Aug 3. PMID 22864529
- [Background] Ito H, Kawaai H, Yamazaki S, Suzuki Y. Maximum opening of the mouth by mouth prop during dental procedures increases the risk of upper airway constriction. Ther Clin Risk Manag. 2010 May 25;6:239-48. doi: 10.2147/tcrm.s10187. PMID 20526442
- [Background] Bingham RM, Proctor LT. Airway management. Pediatr Clin North Am. 2008 Aug;55(4):873-86, ix-x. doi: 10.1016/j.pcl.2008.04.004. PMID 18675024